CLINICAL TRIAL: NCT01611116
Title: A Double-blind, Placebo-controlled, Randomized, Multicenter Phase II Trial to Assess the Efficacy of Temsirolimus Added to Standard Primary Therapy in Elderly Patients With Newly Diagnosed AML
Brief Title: Study With Temsirolimus Added to Standard Chemotherapy for Patients Over 60 Years With Acute Myeloblastic Leukemia
Acronym: TOR-AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Christian Brandts, MD, Study Director, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3066K1-1165
Record Dates: First submitted 2012-05-25; First posted 2012-06-04 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — temsirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium chloride solution 0.9% (Placebo Comparator)
  Interventions: Drug: sodium chloride solution 0.9%
- temsirolimus (Experimental)
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: sodium chloride solution 0.9% — intravenous application added to standard chemotherapy on up to 8 predefined days during the course of study treatment
  Arms: sodium chloride solution 0.9%
Drug: temsirolimus — intravenous application added to standard chemotherapy on up to 16 predefined days during the course of study treatment
  Other Names: Torisel
  Arms: temsirolimus

SUMMARY:
Standard chemotherapy is capable of eliminating most leukemic blasts in acute myeloblastic leukemia (AML), while leukemia-initiating cells are not sufficiently eradicated. As a consequence, refractory disease and relapse frequently occur in AML, especially in elderly patients. The investigators propose that the addition of temsirolimus may improve standard AML chemotherapy. Furthermore, temsirolimus may specifically target the leukemia-initiating cells in AML, thereby reducing the risk of leukemia relapse.

The study's main part is preceded by a open label run-in part, in which optimal temsirolimus dose and schedule for the main part o the study will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML (except APL) according to the FAB classification, including AML evolving from MDS or other hematological diseases and AML after previous cytotoxic therapy or radiation (secondary AML)
* Bone marrow aspirate or biopsy contains ≥ 20% blasts of all nucleated cells or differential blood count must contain ≥ 20% blasts. In AML FAB M6 ≥ 30% of non-erythroid cells in the bone marrow must be leukemic blasts. In AML defined by cytogenetic aberrations the proportion of blasts may be < 20%.
* Age ≥ 61 years
* Informed consent, personally signed and dated to participate in the study
* Willingness of male patients whose sexual partners are women of child-bearing potential (WOCBP), to use an effective form of contraception (pearl index < 1%) during the study and at least 6 months thereafter.

Exclusion Criteria:

* Patients who are not eligible for standard chemotherapy
* Previous treatment for AML, except leukapheresis for patients with hyperleukocytosis (leukocytes > 100,000/µl and / or leukostatic syndrome) or hydroxyurea
* Known central nervous system manifestation of AML
* Cardiac Disease: Heart failure NYHA III° or IV°; active coronary artery disease (MI more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias, defined as: ventricular extrasystoles grade LOWN IV, sustained or non-sustained ventricular tachycardias, and history of ventricular fibrillation / ventricular flutter, unless patient is protected by an internal cardioverter / defibrillator or ventricular arrhythmia was attributable to a myocardial ischemia > 6 months before study entry.
* Chronically impaired renal function (creatinine clearance < 30 ml / min)
* Chronic pulmonary disease with relevant hypoxia
* Inadequate liver function (ALT and AST ≥ 2.5 x ULN) if not caused by leukemic infiltration
* Total bilirubin ≥ 1.2 mg/dL if not caused by leukemic infiltration
* Uncontrolled active infection
* Concurrent malignancies other than AML with an estimated life expectancy of less than two years and requiring therapy
* Known HIV and/or hepatitis C infection
* Evidence or history of CNS disease, including primary or metastatic brain tumors, seizure disorders
* History of organ allograft
* Concomitant treatment with kinase inhibitors, angiogenesis inhibitors, calcineurin inhibitors and Mylotarg
* Serious, non-healing wound, ulcer or bone fracture
* Allergy to study medication or excipients in study medication
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardise compliance with the protocol

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-05; Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
median Event Free Survival (EFS) | participants will be followed for one year after start of study treatment
  Event Free Survival defined as time interval from day 1 of study treatment until treatment failure, relapse from complete remission (CR) or incomplete remission (CRi), or death from any cause, whichever occurs first.
event free survival probability | participants will be followed for one year after start of study treatment
  Event Free Survival defined as time interval from day 1 of study treatment until treatment failure, relapse from complete remission (CR) or incomplete remission (CRi), or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
median Event Free Survival (EFS) of AML patients with different cytogenetic and molecular risk groups | participants will be followed for one year after start of study treatment
rate of early response after the first induction cycle in the temsirolimus and the control group | participants will be followed for one year after start of study treatment
rate of early response of AML patients with different cytogenetic and molecular risk groups | participants will be followed for one year after start of study treatment
Complete Remission (CR) rate in the temsirolimus and the control group | participants will be followed for one year after start of study treatment
CR rate of AML patients with different cytogenetic and molecular risk groups | participants will be followed for one year after start of study treatment
Relapse Free Survival (RFS) of AML patients in the temsirolimus and the control group | participants will be followed for one year after start of study treatment
Relapse Free Survival (RFS) of AML patients with different cytogenetic and molecular risk groups | participants will be followed for one year after start of study treatment
Overall Survival (OS) of all AML patients in the temsirolimus and the control group | participants will be followed for one year after start of study treatment
Overall Survival (OS) of AML patients with different cytogenetic and molecular risk groups | participants will be followed for one year after start of study treatment
rate of molecular remissions in the temsirolimus and the control group | participants will be followed for one year after start of study treatment
Number of adverse events in the temsirolimus and the control group | participants will be followed for one year after start of study treatment
rate of molecular relapse after molecular remission of all AML patients in the temsirolimus and the control group after induction therapy and in the course of the first remission | participants will be followed for one year after start of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Brandts, MD, Study Director — Goethe University
Locations (5):
- Germany (5):
  - Charité University Hospital Berlin, Campus Benjamin Franklin, Berlin
  - University Hospital Dresden, Dresden
  - University Hospital Erlangen, Erlangen
  - University Hospital Frankfurt, Frankfurt am Main
  - University Hospital Münster, Münster

REFERENCES:
- [Result] Posting of Results in EUDRACT Database: https://www.clinicaltrialsregister.eu/ctr-search/trial/2011-002365-37/results
- See also: University Cancer Center Frankfurt — http://www.uct-frankfurt.de
- See also: German Competency Network for Leukemia — http://www.kompetenznetz-leukaemie.de